CLINICAL TRIAL: NCT06873932
Title: Efficacy of Orthodontic Tooth Movement Using Beveled and Conventional Attachments in Aligners: a Randomized Split-Mouth Clinical Trial
Brief Title: Efficacy of Orthodontic Tooth Movement Using Beveled and Conventional Attachments in Aligners
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Neodent (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CC.2024.Attachments
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Malocclusion; Tooth Movement Techniques
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm: Beveled attachments (Experimental): The patients will receive beveled attachments on one side of the jaws
  Interventions: Device: Arm 1: Beveled Attachments
- Rectangular Attachments (Active Comparator): The patients will receive rectangular attachments on one side of the jaws
  Interventions: Device: Conventional Rectangular Attachments

INTERVENTIONS:
Device: Arm 1: Beveled Attachments — Beveled attachments applied to 20 teeth in each subgroup (horizontal, vertical, and rotational movements).
  Arms: Arm: Beveled attachments
Device: Conventional Rectangular Attachments — Conventional rectangular attachments applied to 20 teeth in each subgroup (horizontal, vertical, and rotational movements).
  Arms: Rectangular Attachments

SUMMARY:
The objective of this study is to evaluate the efficacy of tooth movement using beveled attachments and conventional attachments. The sample will be consecutively selected, comprising participants seeking orthodontic treatment in a private dental office within the recruitment period (from ethics committee approval to July 2027). Participants will be selected and randomized using a split-mouth study design. Groups will be divided into rectangular and beveled attachments, each further subdivided into subgroups for horizontal movements (Group H), vertical movements (Group V), and rotations (Group R), with 20 teeth/attachments per group, totaling a sample of 120 teeth/attachments. Digital study models will be obtained before the start of treatment and immediately after its completion. Additionally, clinical intraoral and extraoral photographs will be taken (pre- and post-treatment). Measurements will be collected from the initial and final digital models to determine the magnitude and direction of movements resulting from treatment. Descriptive statistics will be calculated for each type of dental movement evaluated. Paired tests will be conducted due to the split-mouth design. Correlation tests will be applied if necessary.

DETAILED DESCRIPTION:
Participant recruitment will take place after approval by the Research Ethics Committee until July 2027. The consultations will occur in a private clinic in Curitiba - PR, Brazil.

Participants will be selected and randomized according to the split-mouth study design. Teeth on each side will have different attachment configurations to aid orthodontic aligner movements. One side will use rectangular attachments, and the other side will use beveled attachments. Groups will be divided as follows:

Group H: 20 teeth/attachments with horizontal displacements (parallel to the occlusal plane) including tipping or mesio-distal translation - premolars and molars.

Group V: 20 teeth/attachments with vertical displacements (extrusion and intrusion) - incisors.

Group R: 20 teeth/attachments with mesio-distal rotations - canines and premolars.

Digital study models (intraoral scanner) will be obtained before and after treatment. These intraoral scans will be analyzed alongside the planned movement models generated by the orthodontic treatment planning software.

Treatment efficacy will be analyzed using tooth-tracking methodology in Geomagic Control X, measuring the differences between planned and achieved movements and calculating the percentage of achieved orthodontic tooth movement.

Additionally, pre- and post-treatment clinical photographs will be taken:

Intraoral:

Frontal in occlusion; Right and left lateral views in occlusion; Occlusal views of upper and lower arches.

Extraoral:

Frontal with lips at rest; Frontal with a wide smile; Profile with lips at rest. All participants will receive orthodontic aligner treatment supervised by a qualified professional capable of providing relevant care under clinical trial conditions. Diagnosis, movement planning, and therapy monitoring procedures (e.g., aligner replacement frequency) for each individual will be established by the researcher, respecting the manufacturer's specified instructions.

The sample size was 30 participants will be recruited, totaling a sample of 120 teeth/attachments.

Participant satisfaction will be recorded pre-treatment, during follow-up, and post-treatment. In this study, oral health-related quality of life will be assessed through the OHIP-14 (Oral Health Impact Profile-14) questionnaire as a measure of participant satisfaction with the treatment.

Initial and final digital models will be imported using software, where measurements will be taken to identify the magnitude and direction of movements resulting from treatment with different attachment types:

Horizontal displacements (parallel to the occlusal plane) including tipping or mesio-distal translation - premolars and molars.

Vertical displacements (extrusion and intrusion) - incisors. Mesio-distal rotations - canines and premolars.

Descriptive statistics will be calculated for each type of tooth movement evaluated and described by mean, standard deviation, median, quartiles, minimum, and maximum. Paired tests will be conducted due to the split-mouth design. Correlation tests will also be applied if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years) with permanent dentition
* Candidates for aligner-based orthodontic treatment
* Require bilateral tooth movements (e.g., extrusion, intrusion, rotation, tipping, mesiodistal translation)
* Provide written informed consent

Exclusion Criteria:

* Contraindications to aligner use (e.g., manufacturer's guidelines)
* Poor oral hygiene, active periodontal disease, or TMJ disorders
* Allergies to aligner materials (e.g., polyurethane, PETG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of dental movement using beveled and conventional attachments | From enrollment to the end of treatment, not exceeding 24 months.
  Difference between the planned movement and the achieved movement, and the percentage of orthodontic dental movement achieved.

SECONDARY OUTCOMES:
To measure dental movements achieved with the treatment. | From enrollment to the end of treatment, not exceeding 24 months.
  To measure the horizontal, vertical, and rotational dental movements achieved with the treatment
Measure the transverse dental changes achieved. | From enrollment to the end of treatment, not exceeding 24 months.
  Transverse dental changes will be analyzed by comparing pre-treatment and post-treatment digital dental scans.
To assess participant satisfaction throughout the treatment. | From enrollment to the end of treatment, not exceeding 24 months.
  Participant satisfaction will be recorded pre-treatment, during follow-up, and post-treatment. In this study, oral health-related quality of life will be assessed through the OHIP-14 (Oral Health Impact Profile-14) questionnaire as a measure of participant satisfaction with the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Private orthodontic clinic, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No